CLINICAL TRIAL: NCT01812486
Title: Dose De-escalation to the Elective Nodal Sites, the Swallowing Apparatus and Neck Soft Tissues for Head and Neck Cancer: Multi-centre, Randomized Phase III Trial Using Image-guided Intensity-modulated Radiotherapy (IG-IMRT)
Brief Title: Dose De-escalation to the Elective Nodal Sites in Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Dr. Sandra Nuyts, Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S50809
Record Dates: First submitted 2013-03-11; First posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control arm (Active Comparator): NID2Gy = 50 Gy Swallowing apparatus: standard dose
  Interventions: Radiation: standard dose
- Experimental de escalated arm (Experimental): NID2Gy = 40 Gy Swallowing apparatus: Dmax ≤ 60 Gy at 1 cm Dmax ≤ 50 Gy at 1.5 cm from the GTV or PSTB edge
  Interventions: Radiation: dose de escalation

INTERVENTIONS:
Radiation: dose de escalation
  Other Names: IMRT
  Arms: Experimental de escalated arm
Radiation: standard dose
  Arms: control arm

SUMMARY:
A randomized clinical trial was initiated to investigate whether a reduction of the dose to the elective nodal sites and the swallowing apparatus delivered by IMRT would result in a reduction of acute and late side effects without compromising tumor control.

DETAILED DESCRIPTION:
1. Study hypothesis

   Dose de-escalation in the elective nodal sites and off-target regions of the swallowing apparatus delivered by IMRT does reduce overall rate of late dysphagia and neck fibrosis comparing to the standard dose to the elective nodal sites.
2. Primary endpoint

   To estimate the difference in overall rate of late dysphagia and neck fibrosis 1 year after the end of radiotherapy in patients receiving dose de-escalation to the elective nodal sites and off-target regions of the swallowing apparatus applying IMRT.
3. Secondary endpoints

Local, regional and distant control Recurrence and site of recurrence Overall, disease-free and disease-specific survival Acute toxicity Quality of life

ELIGIBILITY:
Inclusion Criteria:

oral cavity, oropharynx, hypopharynx and larynx SCC Histolocervical lymph node metastases of unknown primary cancer Primary unresectable tumor and/or patients refused surgery Stage T2-4; T3-4 N0 Tany N1-3 for laryngeal cancer Karnofsky performance status ≥70% Age ≥ 18 years old

Exclusion Criteria:

Treatment combined with brachytherapy Prior irradiation to the head and neck region History of prior malignancies, except for cured non-melanoma skin cancer, curatively treated in-situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease at least 5 years Distant metastases Pregnant or lactating women Patient unlikely to comply with the protocol, i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-05; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
overall rate of late dysphagia and neck fibrosis | 5 years

SECONDARY OUTCOMES:
locoregional control | 5 years
Quality of life | 5 years
Acute dysphagia | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals UZLeuven, Leuven, Belgium

REFERENCES:
- [Derived] Deschuymer S, Nevens D, Duprez F, Daisne JF, Dok R, Laenen A, Voordeckers M, De Neve W, Nuyts S. Randomized clinical trial on reduction of radiotherapy dose to the elective neck in head and neck squamous cell carcinoma; update of the long-term tumor outcome. Radiother Oncol. 2020 Feb;143:24-29. doi: 10.1016/j.radonc.2020.01.005. Epub 2020 Feb 7. PMID 32044165